CLINICAL TRIAL: NCT04564703
Title: Phase II Study of Iberdomide (Cc220) Maintenance After Autologous Stem Cell Transplantation in Newly Diagnosed Multiple Myeloma Patients
Brief Title: Iberdomide (Cc220) Maintenance After Asct in Newly Diagnosed MM Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting European Myeloma Network (Network)
Collaborators: Healt Data Specialists - HeaDS (CRO) (Unknown); EMN Research Italy Impresa Sociale Srl (Unknown)
Responsible Party: Sponsor
Organization: European Myeloma Network B.V. (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMN26
Record Dates: First submitted 2020-09-14; First posted 2020-09-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
Keywords: Newly diagnosed MM patients; IBERDOMIDE; Maintenance
MeSH Terms: conditions — Multiple Myeloma | interventions — iberdomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cohort 1 (Experimental): Iberdomide will be given orally at 1.3 mg/day, from day 1 to 21 of a 28-day cycle, continuously, until progressive disease (PD) or unacceptable toxicity.
  Interventions: Drug: Iberdomide
- cohort 2 (Experimental): Iberdomide will be given orally at 1.0 mg/day, from day 1 to 21 of a 28-day cycle, continuously, until progressive disease (PD) or unacceptable toxicity.
  Interventions: Drug: Iberdomide
- cohort 3 (Experimental): Iberdomide will be given orally at 0.75 mg/day, from day 1 to 21 of a 28-day cycle, continuously, until progressive disease (PD) or unacceptable toxicity.
  Interventions: Drug: Iberdomide

INTERVENTIONS:
Drug: Iberdomide — IBERDOMIDE (CC220) IN MAINTENANCE AFTER AUTOLOGOUS STEM CELL TRANSPLANTION IN NEWLY DIAGNOSED MULTIPLE MYELOMA PATIENTS

SUMMARY:
This is a phase II study to evaluate the efficacy and safety of different doses of iberdomide continuous therapy as maintenancetreatment after transplant.

DETAILED DESCRIPTION:
This is a phase II study with two parallel cohorts of newly diagnosed multiple myeloma (NDMM) patients in at least partial response (PR) after induction with proteasome inhibitors (PIs) plus IMIDs and single or double ASCT Subjects will receive two dose levels of Iberdomide, they will be evaluated for efficacy and safety. In case, in one cohort will be registered unacceptable toxicity, a third cohort will be opened. Subjects will receive treatment until progression, intolerance or unacceptable toxicity. Subsequently subjects will be followed for 24 months. The maximum number of subjects is 130 for cohort 1 and 2, 160 in case a third cohort will be opened.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with newly diagnosed MM, requiring therapy due to the presence of CRAB symptoms or myeloma defining events and measurable disease (sPEP >0.5 g/dL and/or uPEP > 200 mg/24h and/or FLC involved > 10 mg/dL with abnormal FLC ratio) before induction therapy with a PI and IMID-containing regimen-
* Subjects with complete baseline evaluation at the time of diagnosis according to revised International Staging System (R-ISS) (cytogenetic profile, ISS and LDH)
* Subjects treated with proteasome inhibitor plus immunomodulatory drug-based induction (3-6 cycles), followed by single or double autologous stem cell transplant (ASCT) with melphalan as condItioning regimen +/- consolidation.
* Subjects within 12 months from diagnosis and 120 days after last ASCT, who achieved at least a partial response (PR) after ASCT, according to IMWG criteria
* Subjects willing and able to follow the trial procedures
* Subjects must understand and voluntary sign an ICF prior to any study related assessment/procedurs being conducted
* Age ≥18 years
* ECOG performance status 0-1
* A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months) and must:

  1. Have two negative pregnancy tests as verified by the Investigator prior to starting study treatment. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence* from heterosexual contact.
  2. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with two forms of contraception: one highly effective, and one additional effective (barrier) measure of contraception without interruption 28 days prior to starting investigational product, during the study treatment (including dose interruptions), and for at least 28 days after the last dose of CC-220, 90 days after the last dose of cyclophosphamide, whichever is longer. Contraception requirements are detailed in Appendix H.
* Male subjects must:

  a. Practice true abstinence* (which must be reviewed on a monthly basis and source documented) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 90 days following the last dose of study treatment, even if he has undergone a successful vasectomy.

  * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.]
* Males must agree to refrain from donating sperm while on study treatment, during dose interruptions and for at least 90 days following last dose of study treatment.
* All subjects must agree to refrain from donating blood while on study treatment, during dose interruptions and for at least 28 days following the last dose of study treatment.
* All male and female subjects must follow all requirements defined in the Pregnancy Prevention Program (v5.1). See Appendix I for CC-220 Pregnancy Prevention Plan for Subjects in Clinical Trials.
* Subject agree to refrain from donating blood while on iberdomide, during dose interruption and for at least 28 days following the last iberdomide dose
* Baseline values:

ANC ≥1.0 x 109/L without use of growth factors; PLTs≥75 x109/L (transfusions within 14 days from Day1 cycle 1 to achieve this cut off are not allowed); Hb >8 g/dL (transfusions within 14 days from Day1 cycle 1 to achieve this cut off are not allowed); • Life expectancy ≥ 3 months

Exclusion Criteria:

* • Systemic AL amyloidosis or plasma cell leukemia (>2.0x109/L circulating plasma cells by standard differential) or Waldenstrom's macroglobulinemia

  * Subject has known meningeal involvement of multiple myeloma
  * History of active malignancy during the past 5 years, except squamous cell and basal cell carcinomas of the skin and carcinoma in situ of the cervix or breast and incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) or prostate cancer that is cured, or malignancy that in the opinion of the local investigator, with concurrence with the principal investigator, is considered cured with minimal risk of recurrence within 3 years.
  * Subject with any one of the following: clinically significant abnormal electrocardiogram (ECG) findings at screening; congestive heart failure (New York Heart Association Class III or IV); myocardial infarction within 12 months prior to starting iberdomide; unstable or poorly controlled angina pectoris, including Prinzmetal variant; clinically significant pericardial disease
  * Peripheral neuropathy of ≥grade 2.
  * Subject has any concurrent severe and/or uncontrolled medical condition or psychiatric disease that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study or that confounds the ability to interpret data from the study.
  * Subjects with gastrointestinal disease that may significantly alter the absorption of iberdomide
  * Subject with known history of anaphylaxis or hypersensitivity to thalidomide, lenalidomide, pomalidomide
  * Subject with known or suspected hypersensitivity to excipients contained in the formulation of iberdomide
  * Subjects has current or prior use of immunosuppressive medication within 14 days prior to starting therapy with iberdomide (exceptions are intranasal, inhaled, topical or local steroids injections; systemic corticosteroids at doses not exceeding 10 mg/day of prednisone or equivalent; steroids as premedication for hypersensitivity reactions)
  * Subject has taken a strong inhibitor or inducer of CYP3A4/5 including grapefruit, St John's wort or related products within 2 weeks prior to dosing and during the course of study
  * Subject known to test positive for HIV or have active hepatitis A, B or C
  * Subjects is unable or unwilling to undergo protocol required thromboembolism prophylaxis
  * Subject is a female who is pregnant nursing or breastfeeding or who intends to become pregnant during the participation
  * Baseline lab values:
* Creatinine clearance ≤30 ml/min.
* Significant hepatic dysfunction (total bilirubin > 1.5x ULN or AST/ALT > 2.5x ULN), or > 3.0 mg/dL for subjects with documented Gilbert's syndrome unless related to myeloma
* Corrected serum calcium>13.5 mg/dL (3.4 mmol/L) • Any clinical condition at screening that would preclude subject from completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy: rate of improvement in response with iberdomide maintenance after autologous stem cell transplantation (ASCT) | 6 months of treatment
  Response improvement rate within 6 months will be measured as the number of subjects that improve response according to IMWG criteria (from PR to ≥VGPR; from VGPR to ≥CR; from CR to >sCR) within the end of sixth cycle of treatment.
Rate of dose reductions/discontinuations with iberdomide maintenance after ASCT | 6 months of treatment
  Dose reductions/discontinuation rate within 6 months will be measured as the number of subjects that discontinued treatment or have a dose modification within the end of sixth cycle of treatment

SECONDARY OUTCOMES:
Rate of next-generation flow (NGF ) minimal residual disease (MRD) conversion from positive to negative. | 6 months of treatment
  Rate of NGF Minimal residual disease (MRD) conversion from positive to negative.The MRD conversion rate at 6 months is determined as the proportion of subjects with MRD negativity (*10-5 sensitivity level, by NGF) after 6 months converted from status as Positive at screening.
Rate of next-generation flow (NGF ) minimal residual disease (MRD) conversion from positive to negative. | 12 months of treatment
  The MRD conversion rate at 12 months is determined as the proportion of subjects with MRD negativity (*10-5 sensitivity level, by NGF) after 12 months converted from status as Positive at screening. Subjects who withdraw from the study or are lost to follow up before post 12 months MRD evaluation, the best MRD assessment will be considered
Rate of next-generation flow (NGF ) minimal residual disease (MRD) conversion from positive to negative. | 12 months of treatment
  The best MRD conversion rate within 12 months is determined as the proportion of subjects with MRD negativity (*10-5 sensitivity level, by NGF) within 12 months converted from status as Positive at screening. Subjects who withdraw from the study or are lost to follow up before MRD evaluation, the best MRD assessment will be considered.
Rate of adverse events | approximately 60 months
  The analysis of safety as defined by type, frequency and severity will be done primarily by tabulation of the incidence of AEs as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. In the by-subject analysis, a subject having the same event more than once will be counted only once.
  AEs will be summarized by worst CTCAE grade
Safety in different subset of subjects with different prognostic features | approximately 60 months
  Determine whether rate of adverse events may change in subgroups with different prognosis according to current prognostic factors
Efficacy in different subset of subjects with different prognostic features | approximately 60 months
  Determine whether tumor response in terms of response and survival may change in subgroups with different prognosis according to current prognostic factors
Time to Progression (TTP) | approximately 60 months
  TTP will be measured by protocol from the date of start of therapy and according to ITT from the date of eligibility confirmation to the date of first observation of PD, or deaths for PD. Subjects who have not progressed or who withdraw from the study or die from causes other than PD will be censored at the time of the last disease assessment. Subjects lost to FU will also be censored at the time of last complete disease assessment.
Progression Free Survival (PFS) | approximately 60 months
  PFS will be measured by protocol from the date of start of therapy and according to ITT from the date of eligibility confirmation to the date of first observation of PD, or death from any cause as an event. Subjects who have not progressed or who withdraw from the study or who were lost to FU will be censored at the time of the last disease assessment.
Time to next therapy (TNT) | approximately 60 months
  TNT will be measured by protocol from the date of start of therapy and according to ITT from the date of eligibility confirmation to the date of next anti-myeloma therapy. Death due to any cause before starting therapy will be considered an event. Subjects who have not progressed or who withdraw from the study

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gay, MD, Principal Investigator — University of Torino, Via Nizza 52, 10126 Torino; Niels van De Donk, MD, Principal Investigator — Amsterdam UMC, VU University Medical Center, De Boelelaan 1117, Amsterdam
Locations (4):
- CHU Hôtel-Dieu, 1, place Alexis Ricordeau, 44093 NANTES Cedex 1, FRANCE, Nantes, France
- Alexandra General Hospital -Department of Clinical Therapeutics N.K. Univ. of Athens, Athens, Greece
- Ospedale Generale Regionale-Divisione di Ematologia e Centro Trapianto Midollo Osseo, Bolzano, Italy
- Vrije Universiteit Medical Center (VUMC), Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No